CLINICAL TRIAL: NCT02637531
Title: A Phase 1/1b First-In-Human, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IPI-549 Monotherapy and in Combination With Nivolumab in Subjects With Advanced Solid Tumors
Brief Title: A Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IPI-549
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-549-01
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumors (Part A/B/C/D); Non-small Cell Lung Cancer (Part E); Melanoma (Part E); Squamous Cell Cancer of the Head and Neck (Part E); Triple Negative Breast Cancer (Part F); Adrenocortical Carcinoma (Part G); Mesothelioma (Part G); High-circulating Myeloid-derived Suppressor Cells (Part H)
Keywords: IPI-549; Phase 1; Advanced Solid Tumor; Non-small cell lung cancer; Melanoma; PI3K; Squamous Cell Cancer of the Head and Neck; Triple Negative Breast Cancer; Adrenocortical Carcinoma; Mesothelioma; High-circulating myeloid-derived suppressor cells (MDSCs); eganelisib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Triple Negative Breast Neoplasms; Adrenocortical Carcinoma; Mesothelioma | interventions — IPI-549; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Part A/B: IPI-549 Dose Escalation (Experimental): Participants receive IPI-549 orally (PO) once a day (QD) for Part A and twice a day (BID) in Part B until disease progression.
  Interventions: Drug: IPI-549 (eganelisib)
- Part C: IPI-549 and nivolumab (Experimental): Participants receive IPI-549 (dose determined from Part A/B) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Part D: IPI-549 Monotherapy (Experimental): Participants receive IPI-549 (dose determined from Part A/B) orally until disease progression.
  Interventions: Drug: IPI-549 (eganelisib)
- Part D Annex: IPI-549 and nivolumab (Experimental): Participants receive IPI-549 (dose determined from Part A/B/C) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Part E: NSCLC: IPI-549 and nivolumab (Experimental): Participants with NSCLC receive IPI-549 (dose determined from Part A/B/C) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Part E: Melanoma: IPI-549 and nivolumab (Experimental): Participants with melanoma receive IPI-549 (dose determined from Part A/B/C) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Part E: SCCHN: IPI-549 and nivolumab (Experimental): Participants with squamous cell cancer of the head and neck receive IPI-549 (dose determined from Part A/B/C) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Part F: TNBC: IPI-549 and nivolumab (Experimental): Participants with triple negative breast cancer receive IPI-549 (dose determined from Part A/B/C) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Part G: ACC: IPI-549 and nivolumab (Experimental): Participants with adrenocortical carcinoma receive IPI-549 (dose determined from Part A/B/C) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Part G: Mesothelioma: IPI-549 and nivolumab (Experimental): Participants with mesothelioma receive IPI-549 (dose determined from Part A/B/C) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab
- Part H: High-circulating MDSCs: IPI-549 and nivolumab (Experimental): Participants with high-circulating MDSCs receive IPI-549 (dose determined from Part A/B/C) orally in combination with nivolumab IV infusion (240 mg) every 2 weeks.
  Interventions: Drug: IPI-549 (eganelisib); Drug: Nivolumab

INTERVENTIONS:
Drug: IPI-549 (eganelisib) — IPI-549 daily dose administered orally in 28-day cycles (Part A/BC/D/D-Annex/E)
Drug: Nivolumab — Nivolumab (240 mg, Q2W) administered intravenously (IV) in 28-day cycles (Part C/D-Annex/E).
  Other Names: OPDIVO
  Arms: Part C: IPI-549 and nivolumab; Part D Annex: IPI-549 and nivolumab; Part E: Melanoma: IPI-549 and nivolumab; Part E: NSCLC: IPI-549 and nivolumab; Part E: SCCHN: IPI-549 and nivolumab; Part F: TNBC: IPI-549 and nivolumab; Part G: ACC: IPI-549 and nivolumab; Part G: Mesothelioma: IPI-549 and nivolumab; Part H: High-circulating MDSCs: IPI-549 and nivolumab

SUMMARY:
This dose-escalation study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of IPI-549 monotherapy and IPI-549 in combination with nivolumab in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
Study IPI-549-01 is a first-in-human multicenter, open-label, up to five-part Phase 1/1b dose-escalation study designed to evaluate safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of IPI-549 monotherapy and IPI-549 in combination with nivolumab in subjects with advanced solid tumors.

Approximately 175 subjects will receive IPI-549, either as a monotherapy or in combination with nivolumab. Subjects will receive IPI-549 until the maximum tolerated dose (MTD) is achieved or until disease progression or unacceptable toxicity.

Part A (QD dosing) (and Part B (BID dosing) if necessary) a dose escalation part of the study will evaluate the safety and tolerability, PK, and PD of IPI-549 as a single agent in subjects with advanced solid tumors. Part A/B will determine the recommended phase 2 dose (RP2D) for IPI-549 single agent that is going to be administered in Part D as a single agent and Part C in combination with nivolumab.

Part C a dose-escalation part of the study will evaluate the safety and tolerability, PK, and PD of IPI-549 when administered in combination with IV nivolumab 240 mg every 2 weeks (Q2W) in subjects with advanced solid tumors. Part C will determine the RP2D for the combination of IPI-549 and nivolumab (combination RP2D).

Part D will evaluate the safety, tolerability, PK, PD, and preliminary clinical activity of IPI-549 administered as a single agent in a cohort of subjects with advanced solid tumors. Part D, Cycle 2 will also include a pilot food (a high-fat meal) effect evaluation that will have 8 subjects out of the entire cohort of subjects participating in the Part D.

Part E will evaluate the safety, tolerability, PK, PD, and preliminary clinical activity of IPI-549 in combination with intravenous (IV) nivolumab 240 mg Q2W in a cohort of subjects with non-small cell lung cancer (NSCLC), a cohort of subjects with melanoma and a cohort of subjects with Squamous Cell Cancer of the Head and Neck (SCCHN). One or more cohorts of subjects with additional tumor types may be enrolled if supported by data generated in dose escalation or earlier expansion cohorts. To be eligible for enrollment in Part E, subjects must have received an anti-PD1/PD-L1 as their most recent treatment prior to study entry. The dose level to be administered in Part E will be the combination RP2D as determined in Part C.

Part F will evaluate the safety, tolerability, PK, PD, and preliminary clinical activity of IPI-549 in combination with intravenous (IV) nivolumab 240 mg Q2W in a cohort of subjects with triple negative breast cancer (TNBC). One or more cohorts of subjects with additional tumor types may be enrolled if supported by data generated in dose escalation or earlier expansion cohorts. To be eligible for enrollment in Part E, subjects must have no prior anti-PD1/PD-L1 therapy. The dose level to be administered in Part E will be the combination RP2D as determined in Part C.

Part G will evaluate the safety, tolerability, PK, PD, and preliminary clinical activity of IPI-549 in combination with intravenous (IV) nivolumab 240 mg Q2W in a cohort of subjects with adrenocortical carcinoma (ACC) and a cohort of subjects with mesothelioma who have received at least first line available therapy. One or more cohorts of subjects with additional tumor types may be enrolled if supported by data generated in dose escalation or earlier expansion cohorts. The dose level to be administered in Part E will be the combination RP2D as determined in Part C.

Part H will evaluate the safety, tolerability, PK, and preliminary clinical activity of IPI-549 in combination with IV nivolumab 240 mg Q2W in subjects with advanced cancer with high-circulating MDSCs (ie, ≥ 20.5% as measured by Serametrix CLIA-certified assay); other indication(s) are to be determined. For subject's with a microsatellite instability-high tumor, or tumor type for which anti-PD-1/anti-PD-L1 therapy is considered standard of care, that subject must have previously received an anti-PD-1 or anti-PD-L1 therapy.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet the following criteria for inclusion:

* ≥ 18 years of age
* Life expectancy of ≥ 3 months
* Histological or cytological evidence of advanced and/or metastatic carcinoma or melanoma , excluding sarcoma
* At least 1 measurable disease lesion as defined by RECIST 1.1
* Serum creatinine clearance ≥ 60 mL/min and serum creatinine ≤ 2.0 x the upper limit of normal (ULN) as determined by either of the following: Estimation as calculated by Cockcroft-Gault equation or Direct measurement by 24-hour urine collection
* Total bilirubin ≤ 1.5 x ULN (unless elevated due to Gilbert's syndrome)
* Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 x ULN (<5x ULN if liver metastasis)
* Adequate hematological function, defined as absolute neutrophil count ≥1.5 x 109/L, hemoglobin ≥ 9.0 g/dL, and platelet count ≥ 100 x 109/L
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (corresponds to Karnofsky Performance Status (KPS) ≥ 60%)

Subjects entering Part A, B, C, or D must also meet the following additional criterion:

• Failure to respond to standard therapy, or for whom no appropriate therapies are available (based on the judgement of the Investigator)

Subjects entering Part D, E, F or G must also meet the following additional criterion:

• Willing to undergo 1 pre-treatment and 1 on-treatment tumor biopsy

Subjects entering Part E must also meet the following additional criteria:

* Histological or cytological evidence of NSCLC, melanoma, , human papillomavirus (HPV) positive or HPV negative SCCHN (oral cavity, pharynx, hypopharynx, larynx, nasopharyngeal [including undifferentiated nasopharyngeal carcinoma]), or another tumor type to be determined
* Failure to respond to standard therapy, or for whom no appropriate therapies are available (based on the judgment of the Investigator The most recent treatment prior to study entry must be an anti-PD-1 or anti-PD-L1 antibody given as either monotherapy or in combination
* Subjects with NSCLC Tumors that harbor an actionable genetic alteration for which there is a corresponding approved therapy for that specific alteration (including but not limited to alterations in EGFR, ALK, and ROS) must have progressed on, or had intolerance to, the respective therapy

Subjects entering Part F must also meet the following additional criteria:

* Histological or cytological evidence of estrogen-receptor negative (ER-), progesterone receptor negative (PgR-) and human epidermal growth factor-2 receptor negative (HER2-) Breast Cancer by local laboratory testing, based on last available tumor tissue; or another tumor type to be determined

  * ER/PgR negativity to follow local guidelines
  * If IHC HER2 2+, a negative FISH test is required
  * Inflammatory triple negative breast cancer is allowed
* Must have received and failed/progressed a cytotoxic chemotherapy as first line therapy per standard of care
* No prior anti-PD-1 or anti-PD-L1 therapy

Subjects entering Part G must also meet the following additional criteria:

* Histological or cytological evidence of ACC, mesothelioma, or another tumor type to be determined

  * Both pleural and peritoneal mesothelioma are allowed
  * Epithelioid, sarcomatoid, or biphasic mesothelioma subtypes are allowed
* Progression after at least first line available therapy

Patients entering Part H must also meet the following additional criteria:

High-circulating MDSCs, currently defined for this study as MDSCs

≥ 20.5% as measured by CLIA-certified Serametrix assay Microsatellite status of tumor has been determined Patients with tumors that are microsatellite instability-high must have previously received an anti-PD-1/anti-PD-L1 therapy and progressed on therapy If patient's tumor type is one for which anti-PD-1/anti-PD-L1 therapy is standard of care, patient must have previously received an anti-PD-1 or anti-PD-L1 therapy and progressed while on that therapy

Exclusion Criteria:

Subjects are to be excluded from the study if they meet any of the following criteria:

* Severe allergic or anaphylactic reaction to any monoclonal antibody therapy, murine protein, or known hypersensitivity to any excipient in the study drugs
* Major surgery within 4 weeks prior to Screening
* Subjects who have been treated with chemotherapy, biologic therapy, or other investigational agent within < 5 times the half-life of the agent or < 28 days (whichever is shorter) of starting study drug

NOTE: Subjects whose immediate prior treatment was with nivolumab may start study drug 2 weeks after the last dose of nivolumab

* Symptomatic or untreated brain metastases
* Primary central nervous system (CNS) malignancy
* Infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C virus
* Ongoing treatment with chronic immunosuppressants (eg, cyclosporine) or systemic steroids
* Ongoing systemic bacterial, fungal, or viral infections at Screening

NOTE: Subjects on antimicrobial, antifungal, or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met

* Administration of a live vaccine within 6 weeks of first dose of study drug
* Administration of any of the following within 1 week prior to the administration of study drug:

  * Strong inhibitors or inducers of CYP3A4, including grapefruit products and herbal supplements
  * P-glycoprotein (P-gp) inhibitors
  * Warfarin, phenytoin, or other substrates of CYP2C8 or CYP2C9 with a narrow therapeutic range
  * Medications associated with QTc interval prolongation or Torsades de Pointes
* Baseline QT interval corrected with Fridericia's method (QTcF) > 480 ms (average of triplicate readings) NOTE: criterion does not apply to subjects with a right or left bundle branch block
* Parts C, D-Annex, and E only: Subjects with active, known, or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Prior surgery or gastrointestinal dysfunction that may affect drug absorption (eg, gastric bypass surgery, gastrectomy)
* Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix, or prostate intraepithelial neoplasia
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* History of peptic ulcer and/or gastrointestinal bleed
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to Screening
* Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the subject associated with his or her participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2015-12; Primary Completion 2022-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Part A/B/C: Dose Limiting Toxicities (DLT) | From date of initial dose until up to 28 days for IPI-549
Part D/E: Adverse Events (AE) and safety laboratory values | Number of patients with Clinically significant abnormal laboratory values and adverse events that are related to treatment from date of initial dose until 30 days after last dose of IPI-549 and 100 days after the last dose of Nivolumab

SECONDARY OUTCOMES:
Part A/B: Adverse Events (AE) and safety laboratory values | Number of patients with Clinically significant abnormal laboratory values and adverse events that are related to treatment assessed during every visit for duration of study participation which is estimated to be 24 months
Part A/B: Plasma concentrations of IPI-549 (metabolites, as appropriate) | Assessed during Days 1- 22 of Cycles 1 and 2, Assessed During Day 1 of Cycles 3 and 4
Part A/B: Overall response rate (ORR), complete response/remission (CR) or partial response/remission (PR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part A/B: Duration of response (DoR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part C: Adverse Events (AE) and safety laboratory values | Number of patients with Clinically significant abnormal laboratory values and adverse events that are related to treatment assessed during every visit for duration of study participation which is estimated to be 24 months
Part C: Plasma concentrations of IPI-549 (metabolites as appropriate) | Assessed during Days 1- 2 of Cycles 1 and 2
Part C: Overall Response Rate (ORR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part C: Duration of Response (DoR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part D: Overall Response Rate (ORR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part D: Duration of Response (DoR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part D: Progression-Free Survival (PFS) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part D: Overall Survival (OS) | Estimated to be 3 years
Part D: Plasma concentrations of IPI-549 (and metabolites, as appropriate) | Assessed during Days 1- 15 of Cycles 1 and 2, Assessed During Day 1 of Cycles 3 and 4
Part E:Overall Response Rate (ORR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part F:Overall Response Rate (ORR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part G:Overall Response Rate (ORR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part E: Duration of Response (DoR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part F: Duration of Response (DoR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part G: Duration of Response (DoR) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part E: Progression Free Survival (PFS) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part F: Progression Free Survival (PFS) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part G: Progression Free Survival (PFS) | Responses Assessed in Cycle 3 and every odd cycle through study completion, an average of 1 year
Part E: Overall Survival (OS) | Estimated to be 3 years
Part F: Overall Survival (OS) | Estimated to be 3 years
Part G: Overall Survival (OS) | Estimated to be 3 years
Part E: Plasma concentrations of IPI-549 (and metabolites, as appropriate) | Assessed during Days 1- 2 of Cycles 1 and 2
Part F: Plasma concentrations of IPI-549 (and metabolites, as appropriate) | Assessed during Days 1- 2 of Cycles 1 and 2
Part G: Plasma concentrations of IPI-549 (and metabolites, as appropriate) | Assessed during Days 1- 2 of Cycles 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Feng Chi, MD, Study Director — Infinity Pharmaceutical, Inc.
Locations (11):
- United States (11):
  - UCSD, San Diego, California
  - UCLA, Santa Monica, California
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research and Treatment (START), San Antonio, Texas

REFERENCES:
- [Derived] O'Connell BC, Hubbard C, Zizlsperger N, Fitzgerald D, Kutok JL, Varner J, Ilaria R Jr, Cobleigh MA, Juric D, Tkaczuk KHR, Elias A, Lee A, Dakhil S, Hamilton E, Soliman H, Peluso S. Eganelisib combined with immune checkpoint inhibitor therapy and chemotherapy in frontline metastatic triple-negative breast cancer triggers macrophage reprogramming, immune activation and extracellular matrix reorganization in the tumor microenvironment. J Immunother Cancer. 2024 Aug 30;12(8):e009160. doi: 10.1136/jitc-2024-009160. PMID 39214650